CLINICAL TRIAL: NCT00071474
Title: Shamanic Healing for Women With Temporomandibular Joint Disorders (TMDs)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21AT000951-01A2 (NIH)
Record Dates: First submitted 2003-10-23; First posted 2003-10-24 (Estimated); Last update posted 2007-01-24 (Estimated); Status verified 2007-01

CONDITIONS: Temporomandibular Disorders
Keywords: temporomandibular disroders; shamanism; chronic pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Chronic Pain

INTERVENTIONS:
Procedure: shamanic healing

SUMMARY:
This is a Phase I study to examine the feasibility and safety of shamanic (spiritual) healing for treating temporomandibular joint disorders (TMDs).

DETAILED DESCRIPTION:
Traditional systems of healing, such as shamanism, do not readily lend themselves to conventional research methods, yet studying their effectiveness is especially germane in the case of chronic conditions that involve an emotional component and that elude allopathic treatment regimens. Temporomandibular joint disorders (TMDs), which affect up to 10% of the adult population, are a prime example of such conditions. Traditional treatment outcomes for TMD pain are often unsatisfactory. Moreover, in women age 25-55 (the age-sex group most affected), TMD is often found in association with depression, anxiety, sleep disturbances, gastrointestinal symptoms, frequent infection,and fibromyalgia. Because these multiple and complex symptoms suggest a loss of spirit or life energy, they may be particularly susceptible to treatment by shamanic (spiritual) healing, which aims to bring disturbed physical, mental, and emotional systems into balance. This phase I study will develop methods to evaluate shamanic healing as an intervention for TMD and will evaluate the feasibility of conducting randomized clinical trials of shamanic healing.

ELIGIBILITY:
Inclusion criteria:

* Females Age 25-55
* TMD Research Diagnosis Criteria (RDC) clinical diagnosis of myofacial pain with or without disc displacement, arthralgia, arthritis, or arthosis
* Three or more significant systemic conditions, e.g. depression, fibromyalgia, GI or reproductive disturbances, upper respiratory problems, etc. in the preceding 2 years.

Exclusion criteria:

* Diagnosed organic or medication induced major mental illness (e.g., schizophrenia, bipolar)
* Other neurological diagnoses (epilepsy, Parkinsons)
* Pregnancy

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25
Dates: Start 2003-08; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Vuckovic, MD, Principal Investigator — Center for Health Research, Northwest
Locations (1):
- Center for Health Research, Northwest, Portland, Oregon, United States